CLINICAL TRIAL: NCT05330806
Title: Collagenase Chemonucleolysis vs Percutaneous Endoscopic Lumbar Discectomy (PELD) for Lumbar Disc Herniation, a Randomized Controlled Trial
Brief Title: Collagenase Chemonucleolysis vs Percutaneous Endoscopic Lumbar Discectomy (PELD) for Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ShenzhenPH spine wang05
Record Dates: First submitted 2022-03-24; First posted 2022-04-15 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagenase chemonucleolysis (Experimental): After local anesthesia, and the puncture point was 8-12cm on the side of the paraspinous process under C arm fluoroscopy. The needle was punctured though the skin with an angle of 45-60 to the posterior of the vertebral via "safe" entry zone to the herniated site outside the intervertebral disc under the epidural space. The syringe was drawn back to confirm that no blood or cerebrospinal fluid was flowing out, Contrast agents were injected to make sure no flows out of the spinal canal. 600 unit collagenase was dissolved in 2ml normal saline and injected slowly with rate of 1ml per minute. The needle was removed and keep the dorsal elevated position for 6-8 hours. Keep away from load bear of lumbar for 3 months.
  Interventions: Procedure: Collagenase chemonucleolysis
- Percutaneous endoscopic lumbar discectomy (PELD) (Active Comparator): For L1-L4 segment, percutaneous endoscopic transforaminal discectomy(PETD) will be performed. An 1cm length incision was made at 8-14cm lateral of the paraspinous process, where a needle puncture to the superior articular process of the lower involved vertebrae of the herniated disc. A series of conical rods are to be introduced, subsequently a reamer is to be introduced through the cannula. After removal of the disc herniation, the cannula and endoscope are to be removed. For L5/S1 segment, percutaneous endoscopic interlaminar discectomy(PEID) was performed. An incision of nearly 7 mm was made at the entry point of the skin, and a series of expansion channels were sequentially inserted into the surface of the ligamentum flavum.Then, the ligamentum flavum and soft tissue around it were removed. Then, the tongue of the working cannula was inserted and rotated into the lateral nerve root. Removed the prominent nucleus pulposus by various nucleus pulposus forceps.
  Interventions: Procedure: Percutaneous endoscopic lumbar discectomy (PELD)

INTERVENTIONS:
Procedure: Collagenase chemonucleolysis — After local anesthesia, and the puncture point was 8-12cm on the side of the paraspinous process under C arm fluoroscopy. The needle was punctured though the skin with an angle of 45-60 to the posterior of the vertebral via "safe" entry zone to the herniated site outside the intervertebral disc under the epidural space. The syringe was drawn back to confirm that no blood or cerebrospinal fluid was flowing out, Contrast agents were injected to make sure no flows out of the spinal canal. 600 unit collagenase was dissolved in 2ml normal saline and injected slowly with rate of 1ml per minute. The needle was removed and keep the dorsal elevated position for 6-8 hours. Keep away from load bear of lumbar for 3 months.
  Arms: Collagenase chemonucleolysis
Procedure: Percutaneous endoscopic lumbar discectomy (PELD) — For L1-L4 segment, percutaneous endoscopic transforaminal discectomy(PETD) will be performed. An 1cm length incision was made at 8-14cm lateral of the paraspinous process, where a needle puncture to the superior articular process of the lower involved vertebrae of the herniated disc. A series of conical rods are to be introduced, subsequently a reamer is to be introduced through the cannula. After removal of the disc herniation, the cannula and endoscope are to be removed. For L5/S1 segment, percutaneous endoscopic interlaminar discectomy(PEID) was performed. An incision of nearly 7 mm was made at the entry point of the skin, and a series of expansion channels were sequentially inserted into the surface of the ligamentum flavum.Then, the ligamentum flavum and soft tissue around it were removed. Then, the tongue of the working cannula was inserted and rotated into the lateral nerve root. Removed the prominent nucleus pulposus by various nucleus pulposus forceps.
  Other Names: Percutaneous transforaminal endoscopic discectomy (PTED) for L1-L4 and percutaneous endoscopic interlaminar discectomy(PEID) for L5-S1 lumbar disc herniation
  Arms: Percutaneous endoscopic lumbar discectomy (PELD)

SUMMARY:
Lumbar disc herniation compressed the nerve cause pain, numbness, weak legs called sciatica, which seriously decrease the quality of life and work efficiency. Both collagenase chemonucleolysis(CCNL) and percutaneous endoscopic lumbar discectomy (PELD) was effective to treat lumbar disc herniation(LDH) requires surgery. whether functional clinical outcomes of CCNL vs PELD effect on LDH was superior, and no study provided convincing evidence.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a common disease with an incidence of 1%-3%, usually manifested as low back pain radiating to the lower extremities, which seriously affects patients' quality of life. Collagen hydrolysis was effective in treating LDH, it makes the protrusion smaller or disappeared, relieving or resolving the compression of nerve root by the protrusion.Percutaneous endoscopic lumbar discectomy (PELD) is a less invasive techniques to treat LDH. However, the outcomes of collagen hydrolysis vs PELD effect was still unknown.

ELIGIBILITY:
Inclusion Criteria:

* at least six weeks of excessive radiating leg pain with no tendency for any clinical improvement despite conservative therapy
* have a nerve root compression by a lumbar disc herniation proven by magnetic resonance imaging

Exclusion Criteria:

* previous surgery at the same or adjacent disc level;
* isthmic or degenerative spondylolisthesis
* pregnancy
* severe comorbid medical or psychiatric disorder (American Society of Anesthesiologists' classification >2);
* severe caudal or cranial sequestration of disc fragments, defined as sequestration towards more than half of the adjacent vertebra;
* contraindication for surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-06-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale/Score of leg | up to 12 months
  Visual Analogue Scale pain assess for leg. Use a ruler about 10cm long, one side is marked with "0" and the other "10" respectively. A score of 0 indicates no pain, 10 indicates the most unbearable pain.
Visual Analogue Scale/Score of lumbar | up to 12 months
  Visual Analogue Scale pain assess for lumbar. Use a ruler about 10cm long, one side is marked with "0" and the other "10" respectively. A score of 0 indicates no pain, 10 indicates the most unbearable pain.
Recurrence rate | up to 12 months
  The percentage of disc herniation recurrence appearance. 0 represents the minimum and 100% represents the maximum.
reoperation | up to 12 months
  The percentage of reoperation rate. 0 represents the minimum and 100% represents the maximum.

SECONDARY OUTCOMES:
The Roland-Morris Disability Questionnaire | up to 12 month
  The Roland-Morris Disability Questionnaire is a health status measure designed to be completed by patients to assess physical disability due to low back pain. The lowest score is 0, the highest 24. The higher the score, the more severe the dysfunction.
the EuroQoL-5D (EQ-5D) | up to 12 month
  EQ-5D descriptive system is a preference-based Health-related quality of life measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. From this, a quality of life score can be calculated ranging from -0.594, indicating a health state worse than death where 0 is death, to 1, indicating full health
Duration of operation | up to 12 month
  Duration of operation time： The minimum value is 1 minute, and the maximum value is 120 minutes
Length of stay in the hospital | up to 12 month
  Length of stay in the hospital： The minimum value is 1 day. The maximum value is 30 days
Major complications | up to 12 month
  Major complications includes cerebrospinal fluid leakage,deep venous thrombosis in the leg, transient increase in neurological deficit, repeated surgery,Opioid analgesics
hospital fees | up to 12 month
  hospital fees ：Minimum 500 yuan, maximum 30,000 yuan
the Oswestry Disability Index (ODI) | up to 12 month
  Disability was evaluated using the Oswestry Disability Index (ODI)
the Medical Outcomes Study 12-item short-form health survey (SF-12) scale | up to 12 month
  SF-12 including mental and physical components, was shorter versions of 36-item Short-Form Health Survey (SF-36) to evaluate life quality
modified MacNab | up to 12 month
  modified MacNab criteria is patient satisfaction with excellent outcomes, good, fair, and poor.
cost-effectiveness | up to 12 month
  Incremental cost-effectiveness ratios (ICERs) will be calculated by dividing the difference in costs by the difference in effects.

CONTACTS AND LOCATIONS:
Overall Officials: Songlin Peng, Doctor, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- ShenzhenPH, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson JN, Cowie JG, Iprenburg M. Transforaminal endoscopic spinal surgery: the future 'gold standard' for discectomy? - A review. Surgeon. 2012 Oct;10(5):290-6. doi: 10.1016/j.surge.2012.05.001. Epub 2012 Jun 15. PMID 22705355
- [Background] Yuan P, Shi X, Wei X, Wang Z, Mu J, Zhang H. Development process and clinical application of collagenase chemonucleolysis in the treatment of lumbar disc herniation: a narrative review in China. Postgrad Med J. 2022 Mar 14:postgradmedj-2021-141208. doi: 10.1136/postgradmedj-2021-141208. Online ahead of print. PMID 35288448
- [Background] Gadjradj PS, Harhangi BS. Percutaneous Transforaminal Endoscopic Discectomy for Lumbar Disk Herniation. Clin Spine Surg. 2016 Nov;29(9):368-371. doi: 10.1097/BSD.0000000000000366. PMID 26945128